CLINICAL TRIAL: NCT03832335
Title: Can we Measure Aniseikonia Tolerance in a Normal Population
Brief Title: A New Measurement of Anseikonia Tolerance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Therese Krarup, Principal investigator, Glostrup University Hospital, Copenhagen
Other Study IDs: 04127
Record Dates: First submitted 2019-01-31; First posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Aniseikonia; Anisometropia and Aniseikonia
MeSH Terms: conditions — Aniseikonia; Anisometropia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phakic group: 21 eyehealthy individuals examined for baseline stereopsis and impact of aniseikonia on stereopsis. An non-invasive measurement.
  Interventions: Diagnostic Test: Measurement of aniseikonia tolerance
- Cataract group: 11 patients awaiting cataract surgery on both eyes. Measurement of baseline stereopsis and impact of artificial induced aniseikonia on stereopsis. A non invasive measurement that are repeated after dilatation of the eyes and again six weeks after surgery.
  Interventions: Diagnostic Test: Measurement of aniseikonia tolerance

INTERVENTIONS:
Diagnostic Test: Measurement of aniseikonia tolerance — Adding sizeglasses of different percent before right and left eye and measure the impact on stereopsis

SUMMARY:
Population 1:

Measure the effect of size glasses from1-9% on stereopsis

Population 2:

Measure the effect of size glasses from 1-9% on stereopsis in two settings:

* before and after cataract surgery
* after dilation of the eye

DETAILED DESCRIPTION:
Population 1:

21 eye healthy phakic individuals. Measurements: baseline stereopsis and stereopsis after size glass (1-9%) is added in front of the right eye and in front og the left eye. This measurement provides details on how much size difference a person can endure without impairing stereopsis.

Population 2:

11 phakic eye healthy individuals awaiting cataract operation on both eyes. Measurements are the same as population 1 but this study group is also measured after dilating the eyes. This is to see if accommodation affects the measurement. A postoperative measurement six weeks after cataract operation is also performed to examine if cataract operation affects the measurement.

ELIGIBILITY:
Inclusion Criteria:

* No previous eye history
* cataract grade <= 1
* visual acuity above 0.8

Exclusion Criteria:

* lack of cooperation
* amblyopia
* axial anisometropia
* ametropia

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: group 1: eyehealthy pahkic individuls group 2: eyehalthy phakic patients awainting cataratc surgery
Sampling Method: Non-Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2019-08-02 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Aniseikonia tolerance | baseline
  How many percent aniseikonia is tolerated before stereopsis is impaired. Measured by first measuring baseline stereopsis and here after adding aniseikonic (size glass) from 1-9% in front of the right and left eye to measure if stereopsis is impaired. If stereopsis is impaired at 4% sizeglas then aniseikonia tolerance is 4%.
Change of Aniseikonia tolerance after surgery | six weeks after surgery
  Measurement of aniseikonia tolerance before and after surgery. Measurement: before and after surgery stereopsis is measured, hereafter aniseikonic glasses (size glass) from 1-9% is added in front of the right and left eye to see if stereopsis is impaired. If stereopsis is impaired with 3% aniseikonic glass then the tolerance is 3%. After surgery the measurement is repeated to examine if the aniseikonia tolerance is the same.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet-glostrup, Glostrup Municipality, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No